CLINICAL TRIAL: NCT05622448
Title: Patient Centered Outcomes and Marginal Bone Changes in CAD/CAM Metallic and Poly Ether Ether Ketone (PEEK) Partial Denture Frameworks
Brief Title: Patient Centered Outcomes and Marginal Bone Changes in CAD/CAM Metallic and (PEEK) Partial Denture Frameworks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Arwa Sedky Abd El-lateef, doctor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: patient satisfaction and RPD
Record Dates: First submitted 2019-07-18; First posted 2022-11-18 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2022-11

CONDITIONS: Patient Satisfaction
Keywords: peek framework; co-cr framework; removable partial denture
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RPD with metallic framework (Active Comparator): removable partial denture with cobalt chromium framework
  Interventions: Other: RPD with PEEK framework; Other: RPD with metallic framework
- RPD with PEEK framework (Experimental): removable partial denture with poly ether ether ketone framework
  Interventions: Other: RPD with PEEK framework; Other: RPD with metallic framework

INTERVENTIONS:
Other: RPD with PEEK framework — removable partial denture with CAD designed PEEK framework
Other: RPD with metallic framework — removable partial denture with cobalt chromium framework

SUMMARY:
To compare PEEK to metallic partial denture frameworks in restoring mandibular Kennedy class I regarding patient satisfaction.

DETAILED DESCRIPTION:
The traditional RPDs with cobalt chromium frameworks and clasps have been proven to be inexpensive, accurate, durable and resistant to distortion .2 On the other hand, they have; unesthetic display of metallic clasps, increased weight, and may provoke an allergic reaction. Because of those drawbacks new metal-free materials have been reported as a replacement of metal alloys in manufacturing RPDs, including; high performance polymers such as polyethylene glycol, polyetherketonketon (PEKK), polyaryletherketone (PAEK) and Polyetheretherketon (PEEK).

Using PEEK and modified PEEK (BioHPP) frameworks were claimed to reduce the distal torqueing and stresses on the abutments in kennedy class I PPDs which is thought to be beneficial for periodontal health of the abutments.10 One of the factors for the dissatisfaction related to the dentures may be attributed to the level of oral perception of each patient. The satisfaction level of the patient is influenced by several factors, including the dentures quality and the plated area, the quality of interaction in the patient-dentist relationship, past experiences with full dentures, and the psychological personality6. In harmony, such factors may promote the improvement of the mastication, the speech, and the aesthetics of the teeth, besides producing less discomfort and pain sensitivity, favoring the comminution of harder food7. However, there are no clinical trials evaluating the effect of PEEK on patient satisfaction and the marginal bone loss around the abutments.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with bilateral free end saddles in the mandible (kennedy class I) with last standing abutment premolar.
2. Opposing dentition is fully intact or restored.
3. Sufficient inter-arch space.
4. Angle's class I maxilla-mandibular relationship.

Exclusion Criteria:

1. Periodontal affection of the abutment teeth.
2. Skeletal mal-relation.
3. Unmotivated patients to maintain adequate oral hygiene to follow up.
4. Patients with neuromuscular and Psychiatric disorders.
5. Systematic disease affecting bone and periodontal health.
6. Insufficient inter-arch space.
7. Patients with physical reasons that could affect follow up.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
patient satisfaction | From enrollment to the last follow up
  Patient satisfaction will be measured using a valid and reliable questionnaire which is Patient satisfaction with lower removable denture questionnaire SLRD-Q.
  likert scale ranges from very good (1) to good (2), neither good nor bad (3), bad (4), and extremely bad (5)
Oral Health Related quality of life | From enrollment to the last follow up

SECONDARY OUTCOMES:
Marginal bone changes. | 2 years
  Radiographic follow up will be performed for marginal bone changes.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No